CLINICAL TRIAL: NCT02173886
Title: A Comparison of Sustained and Extended Release Bupropion Following Bariatric Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: North Dakota State University (Other)
Collaborators: Neuropsychiatric Research Institute, Fargo, North Dakota (Other)
Responsible Party: Principal Investigator, Kristine Steffen, Associate Professor, North Dakota State University
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: BUP; EPSCOR (Other: North Dakota State University)
Record Dates: First submitted 2014-06-19; First posted 2014-06-25 (Estimated); Last update posted 2016-09-28 (Estimated); Status verified 2016-09

CONDITIONS: Roux en Y Gastric Bypass

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bupropion (Experimental): Bupropion SR and XL, single dosages of each separated by a wash-out period
  Interventions: Drug: Bupropion SR and XL

INTERVENTIONS:
Drug: Bupropion SR and XL

SUMMARY:
This study is being conducted to evaluate how the body absorbs and processes the sustained release (SR) and extended release (XL) medication bupropion (Wellbutrin®). Subject who are 1-3 years post gastric bypass surgery will be invited to participate. Non-surgical controls will also be enrolled based on a matching criteria to post gastric bypass subjects. Participants will be asked to complete two 12-hour study days approximately 11 days apart.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female
2. Age 18-65 (inclusive, at time of informed consent)
3. No tobacco use in the past three months.
4. Underwent Roux-en-Y Gastric Bypass weight loss surgery 12-36 months prior to study OR has not had a weight loss surgery but matches the gastric bypass patients on age, gender, and BMI.
5. Ability to read, write and understand English

Exclusion Criteria:

1. Taking a medication that has a clinically significant interaction with bupropion or an interaction that may alter the study data.
2. Hypersensitivity to bupropion or any excipient contained within the dosage forms.
3. Inability to tolerate repeated blood draws.
4. Any history of bipoloar disorder or a psychotic disorder.
5. Current major depressive disorder or current suicidality.
6. Alcohol or substance dependence in the past year.
7. Currently pregnant or lactating or unwillingness to use medically accepted contraception during study
8. Taking a medication which significantly alters gastrointesinal transit time or significantly reduces acid secretion (e.g. routine use of proton pump inhibitors, H2 antagonists, sucralfate).
9. Medical conditon which may increase participant risk with bupropion (e.g., history of significant head injury, seizure disorder, etc.)
10. Self reported history of viral hepatits or HIV.
11. Positive urine drug screen unless documented prescription of a non-interacting medication.
12. History of seizures or epilepsy or other conditions which may increase seizure risk with bupropion as described in the package insert (e.g. history of significant head injury, alcoholism, etc).
13. History of eating disorder such as anorexia nervosa or bulimia.
14. Renal impairment as evidenced by an estimated glomerular filtration rate of less than 60 ml/min/1.73 m2 as reported by the laboratory, or any other abnormality on a renal panel that the medical provider feels puts the participant at risk or may compromise the study data
15. Hepatic insufficiency as defined by any hepatic enzyme greater than 3x the upper limit of normal or other hepatic laboratory abnormalities at the discretion of the medical provider.
16. Any significant electrolyte abnormality on a basic metabolic panel that the medical provider feels may put the subject at risk of a seizure from bupropion.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-06; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Bupropion Plasma Concentrations/Area-Under-the-Curve (AUC) | 48 hours intervals
  The primary aim of this research is to provide a comparison of pharmacokinetic measures associated with a single dose of bupropion SR (sustained release) and bupropion XL (extended release) in Roux-en-Y Gastric Bypass and matched nonsurgical "control" subjects. Comparisons will be based upon bupropion plasma concentrations obtained during the 48 hour sample collection window.

SECONDARY OUTCOMES:
Secondary PK Characteristics | 48 hour collection
  We will also evaluate other PK characteristics associated with bupropion, such as Cmax, Tmax, t1/2, and the ratio of bupropion to the active metabolite ODV, and others.

CONTACTS AND LOCATIONS:
Locations (1):
- Neuropsychiatric Research Institute, Fargo, North Dakota, United States